CLINICAL TRIAL: NCT07013149
Title: ACTION - The Impact of ERA Switching on Risk Stratification in Pulmonary Arterial Hypertension
Brief Title: The Impact of ERA Switching on Risk Stratification in Pulmonary Arterial Hypertension
Acronym: ACTION
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Caio Júlio César dos Santos Fernandes, PhD, University of Sao Paulo General Hospital
Other Study IDs: SGP26691
Record Dates: First submitted 2025-05-14; First posted 2025-06-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension; Pulmonary Arterial Hypertension (PAH); Pulmonary Arterial Hypertension (PAH) (WHO Group 1 PH)
Keywords: Pulmonary Arterial Hypertension; PAH; Endothelin Receptor Antagonists; ERA; Ambrisentan; Bosentan; Drug Switching; Risk Stratification
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who switched from Ambrisentan to Bosentan: This cohort includes adult patients (≥18 years) with a confirmed diagnosis of pulmonary arterial hypertension (PAH) by right heart catheterization who underwent a therapeutic transition from ambrisentan 10 mg once daily to bosentan 125 mg twice daily within the past 6 months. Patients are followed during routine clinical care and assessed between 3 and 6 months after the switch to evaluate changes in risk stratification scores (COMPERA 2.0 and REVEAL Lite 2.0), functional capacity, laboratory parameters, and adverse events. No investigational drug or additional intervention is administered beyond standard care.
  Interventions: Other: Switch from Ambrisentan to Bosentan

INTERVENTIONS:
Other: Switch from Ambrisentan to Bosentan — This intervention refers to a therapeutic switch from ambrisentan (10 mg once daily) to bosentan (125 mg twice daily) in adult patients with pulmonary arterial hypertension (PAH), performed as part of routine clinical care. The switch was not assigned by the investigators but was made based on clinical indications prior to study enrollment. Patients are followed prospectively for up to 6 months to assess changes in risk stratification, functional status, laboratory parameters, and safety outcomes.

SUMMARY:
Pulmonary arterial hypertension (PAH) is a rare, progressive, and potentially fatal disease characterized by increased pulmonary vascular resistance and right ventricular dysfunction. Among the four major molecular pathways involved in PAH pathophysiology-nitric oxide, prostacyclin, activin, and endothelin-1 (ET-1)-the endothelin pathway plays a central role. Endothelin-1 acts on ETA and ETB receptors, inducing vasoconstriction and vascular remodeling.

Endothelin receptor antagonists (ERAs) are cornerstone therapies in PAH. Ambrisentan is selective for ETA and associated with a lower risk of hepatotoxicity. Bosentan, a dual ERA (ETA/ETB), has well-established efficacy but a higher incidence of liver enzyme elevation, with approximately 9% of patients experiencing hepatic side effects and about 2% discontinuing therapy due to hepatotoxicity.

While transitions between ERAs occur in routine clinical practice, data on their clinical impact are scarce. This prospective, observational, single-center cohort study aims to evaluate the effect of switching from ambrisentan to bosentan on risk stratification using the COMPERA 2.0 and REVEAL Lite 2.0 scores at 3-6 months post-switch.

Secondary outcomes include variations in functional class (WHO/NYHA), 6-minute walk distance (6MWD), NT-proBNP levels, incidence of adverse events (with a focus on hepatotoxicity), and hematologic parameters such as anemia.

The study will enroll adult patients (≥18 years) with confirmed PAH by right heart catheterization who have undergone a documented switch from ambrisentan 10 mg to bosentan 125 mg within the last 6 months. The primary endpoint is the proportion of patients whose risk category changes post-transition according to COMPERA 2.0 and REVEAL Lite 2.0. The results are expected to provide clinically relevant insights into therapeutic decisions involving ERA transitions in PAH management.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a progressive, life-threatening disease characterized by pulmonary vascular remodeling, increased pulmonary vascular resistance, and right ventricular failure. Among the key molecular pathways implicated in its pathogenesis, the endothelin system plays a central role. Endothelin-1 (ET-1) promotes vasoconstriction and proliferation primarily through ETA receptors, while ETB receptors help mediate ET-1 clearance and vasodilation.

Endothelin receptor antagonists (ERAs) have become foundational in PAH therapy. Ambrisentan, a selective ETA receptor antagonist, is associated with favorable safety and convenience profiles, including once-daily dosing and lower hepatotoxicity risk. Bosentan, a dual ETA/ETB antagonist, is effective but necessitates regular liver function monitoring due to its known hepatic adverse effects.

In clinical practice, transitioning between ERAs is not uncommon and may be driven by clinical response, side effect profiles, or drug availability. However, limited prospective data exist regarding the safety and clinical implications of switching from ambrisentan to bosentan. Most available evidence is derived from small retrospective cohorts, such as the study by Gong et al. (2022), which suggested that such a transition does not negatively impact hemodynamics, functional class, or exercise capacity.

The ACTION study is a prospective observational cohort designed to systematically evaluate the real-world impact of this therapeutic transition. Specifically, it will assess whether switching from ambrisentan to bosentan influences validated multidimensional risk stratification tools-COMPERA 2.0 and REVEAL Lite 2.0-which integrate clinical, functional, and biochemical parameters to estimate prognosis in PAH patients.

Eligible patients will be adults with confirmed PAH who transitioned therapies within the past six months. Baseline data collected at the time of the medication switch will be compared with follow-up data after 3-6 months of treatment with bosentan. By focusing on risk reclassification, the study aims to determine whether ERA switching introduces measurable clinical impact as captured by these scores.

The study also seeks to capture data on tolerability and laboratory safety, especially related to hepatic enzymes and hematologic changes. Given the absence of randomized data in this area, the ACTION study may provide practical insights into treatment adaptation strategies in PAH, especially in resource-limited settings or when access to specific medications is restricted.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosis of pulmonary arterial hypertension (PAH) by right heart catheterization
* Documented therapeutic switch from ambrisentan (10 mg once daily) to bosentan (125 mg twice daily) within the previous 6 months

Exclusion Criteria:

* History of severe hepatic impairment
* Incomplete clinical or laboratory records that prevent risk score calculation
* Inability to attend clinical follow-up between 3 and 6 months after medication switch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients (≥18 years old) diagnosed with pulmonary arterial hypertension (PAH), confirmed by right heart catheterization, who have undergone a clinically indicated therapeutic switch from ambrisentan to bosentan within the past 6 months. The cohort is representative of a real-world PAH population receiving care at a specialized pulmonary hypertension center. Patients will be prospectively followed for clinical, functional, and laboratory outcomes under routine care conditions.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in risk category according to used scores | 3 to 6 months after Endotelin Receptor Antagonist switch
  Proportion of patients who change their clinical risk category (improvement, worsening, or no change) based on scores between baseline (at the time of medication switch) and follow-up (3 to 6 months after the switch from ambrisentan to bosentan).

SECONDARY OUTCOMES:
Change in Functional Class | 3 to 6 months after Endotelin Receptor Antagonist switch
  Change in functional class between baseline and follow-up (classified as improvement, worsening, or no change), as an indicator of clinical status and exercise tolerance.
Change in 6-Minute Walk Distance (6MWD) | 3 to 6 months after ERA switch
  Change in the distance walked during the 6-minute walk test (6MWD) between baseline and follow-up, measured in meters, to assess exercise capacity.
Change in NT-proBNP Levels | 3 to 6 months after ERA switch
  Variation in serum NT-proBNP levels between baseline and follow-up to assess cardiac stress and right ventricular function.
Incidence of Hepatotoxicity | 3 to 6 months after ERA switch
  Number and proportion of patients who develop elevation of AST or ALT above 3 times the upper limit of normal during the follow-up period, indicating possible liver toxicity.
Change in Hemoglobin Levels | 3 to 6 months after ERA switch
  Change in hemoglobin levels between baseline and follow-up, with specific attention to new or worsening anemia potentially associated with the medication switch.
Change in Individual Parameters of risk stratification | 3 to 6 months after Endotelin Receptor Antagonist switch
  Isolated variation in the individual components of the risk stratification without reclassification into composite risk strata.

CONTACTS AND LOCATIONS:
Locations (1):
- InCor - FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No